CLINICAL TRIAL: NCT02286401
Title: Functional Assessment of Coronary Artery Disease by CTA Flow Encoding
Status: Terminated | Type: Observational
Why Stopped: Recruitment lagged behind goal;exhaustion of funding.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00091805
Record Dates: First submitted 2014-11-03; First posted 2014-11-07 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Coronary Artery Disease
Keywords: myocardial perfusion; coronary atherosclerosis; coronary blood flow; fractional flow reserve; coronary flow reserve
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this pilot study proposal is to test the ability of Transluminal Flow Encoding (TAFE) to evaluate vessel specific ischemia in patients with a clinical indication for invasive coronary angiography (ICA) with fractional flow reserve (FFR) measurements for suspected coronary disease.

DETAILED DESCRIPTION:
The purpose of this pilot study is to test the ability of Transluminal Flow Encoding (TAFE) to evaluate vessel specific ischemia in patients with a clinical indication for invasive coronary angiography (ICA) with fractional flow reserve (FFR) measurements for suspected coronary disease. TAFE is a novel method that derives coronary blood flow from easily obtainable non-invasive coronary CT angiograms.

Participants will undergo a rest coronary CTA, a regadenoson stress CT, and a clinically indicated invasive coronary angiogram. The study aims to determine the accuracy of TAFE compared to invasive fractional flow reserve.

We hypothesize that TAFE-derived coronary blood flow, coronary flow reserve, and myocardial CT perfusion imaging can accurately diagnose an abnormal FFR (<0.80) measured in vessels in patients undergoing invasive coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria A. Male or female patients, age 40 years and older. Women of child bearing potential must demonstrate a negative pregnancy test within 24 hours of the study CT.

B. Referral for invasive coronary angiography for a suspicion of coronary artery disease with possible percutaneous intervention planned.

C. Able to understand and willing to sign the Informed Consent Form.

Exclusion Criteria:

A. Patients with a known history of coronary artery bypass surgery. B. Current or previous ST elevation myocardial infarction (MI), prior MI (confirmed by persistent pathologic Q waves on ECG, clinical reports of CPK-MB or Troponin > three times the upper limit of normal or a fixed perfusion defect on nuclear imaging) C. Current evidence of acute myocardial ischemia, unstable angina, or cardiovascular instability including troponin > than the limit of detection (≥0.06 ng/ml), new ST depression > 1 mm, hypotension with a systolic pressure <90 mm Hg.

D. Known allergy to iodinated contrast media

E. Known or suspected intolerance or contraindication to beta-blockers including:

1. Known allergy to beta-blockers
2. History of moderate to severe bronchospastic lung disease (including moderate to severe asthma) F. Known allergy to regadenoson or aminophylline. G. Any patient not deemed medically stable by a physician. F. Known or suspected severe symptomatic aortic stenosis. G. Severe hypertrophic obstructive cardiomyopathy. H. Evidence of severe symptomatic heart failure (NYHA Class III or IV) at the time of the scan.

I. Inability to lie flat. J. Atrial fibrillation or uncontrolled tachyarrhythmia, or advanced atrioventricular block (second or third degree heart block) K. Elevated serum creatinine (> 1.5mg/dl) OR calculated creatinine clearance of < 60 ml/min (using the Cockcroft-Gault formula) L. History of contrast-induced nephropathy M. Severe pulmonary disease or other disorder that does not allow patient to hold breath for 10 seconds or more.

N. History of organ transplantation O. Acute myocarditis or pericarditis. P. Recent history of illicit drug use (past 3 months) Q. Recent use of dipyridamole containing medications. R. Current pregnancy.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptoms suspicious for obstructive coronary artery disease who will undergo cardiac catheterization.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Coronary Computed Tomography Angiography (CTA), myocardial CT perfusion and TAFE to predict invasive FFR | 2 years
  We will test the diagnostic accuracy of Coronary CTA, myocardial CT perfusion, and transluminal attenuation flow encoding (TAFE) to predict fractional flow reserve (FFR). Coronary CTA and myocardial CT perfusion results will be dichotomous, either normal or abnormal. Coronary CTA will be defined as abnormal when there is a > or = 50% diameter stenosis in a coronary vessel. Myocardial CT perfusion will be defined as abnormal when there is a visually determined myocardial perfusion deficit. TAFE will be a continuous variable in units of ml/min.
  The reference standard will be invasive fractional flow reserve (FFR). FFR will be defined as abnormal when it is less than 0.80.

SECONDARY OUTCOMES:
Diagnostic Accuracy of TAFE-derived coronary blood flow to predict invasive FFR | 2 years
  We will test the diagnostic accuracy of TAFE derived coronary blood flow in ml/min to predict and abnormal FFR (<0.80)

CONTACTS AND LOCATIONS:
Overall Officials: Armin R Zadeh, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States